CLINICAL TRIAL: NCT02704429
Title: An Open-Label, Phase 2, Pilot Study Investigating the Safety, Clinical Activity, Pharmacokinetics, and Pharmacodynamics of Oral Treatment With the BTK Inhibitor PRN1008 in Patients With Newly Diagnosed or Relapsing Pemphigus Vulgaris
Brief Title: A Study of PRN1008 in Adult Patients With Pemphigus Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Principia Biopharma, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRN1008-005; 2015-003564-37 (EudraCT Number)
Record Dates: First submitted 2016-02-24; First posted 2016-03-10 (Estimated); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-12

CONDITIONS: Pemphigus Vulgaris
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Intervention Model Description: Part A with 12 weeks treatment and 12 weeks follow-up. Part B with 24 weeks treatment and 4 weeks follow-up.
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: Yes

ARMS (1):
- PRN1008 (Experimental): Part A: Open-label PRN1008, 12 weeks; 12 weeks follow-up; Part B: Open-label PRN1008, 24 weeks; 4 weeks follow-up
  Interventions: Drug: PRN1008

INTERVENTIONS:
Drug: PRN1008 — Part A dosing was initiated administering 400 mg BID. Intrapatient dose adjustments (reductions and increases) were permitted based upon tolerability and clinical response with the maximum dose allowed up to 600 mg BID for 12 weeks.
  Part B initial dosing was 400 mg QD for 2 weeks with dose escalation to 400 mg BID at the discretion of the Investigator for the purposes of investigating dose response and identifying the minimal efficacious dose of rilzabrutinib for 24 weeks.
  Other Names: BTK inhibitor; Rilzabrutinib

SUMMARY:
Open-label cohort study in adult patients with newly diagnosed or relapsing pemphigus vulgaris, with intra-patient dose-adjustment based on clinical response and BTK occupancy, and with conventional immunosuppressive "rescue treatment", if indicated. The duration of therapy in Part A will be 12 weeks, followed by 12 weeks of follow up. The extension phase, Part B includes 24 weeks of therapy, followed by 4 weeks of follow-up.

DETAILED DESCRIPTION:
Primary Objectives:

To evaluate the safety of PRN1008 in patients with pemphigus vulgaris (PV)

To evaluate the clinical activity of PRN1008 in patients with PV, per criteria in the European Academy of Dermatology and Venereology (EADV) 2014 Pemphigus S2 Guideline (Hertl et al. 2015)

Secondary Objectives

To evaluate the pharmacokinetics (PK) and the pharmacodynamics (PD) of multiple doses of PRN1008 in patients with PV

To evaluate the relationship of PK and PD to each other and to efficacy and safety in this patient population

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged 18 to 80 years old, with biopsy-proven, mild-moderate PV (PDAI 8 to 45) in Part A and mild to severe PV in Part B (PDAI 8 to 60) that are either:

  * newly diagnosed patients (i.e. naïve to an effective induction treatment regimen) for whom an initial period of PRN1008 monotherapy is judged clinically acceptable, or
  * relapsing patients, for whom an initial period of PRN1008 monotherapy, or combination therapy with any of low dose corticosteroid, ie.0.5 mg/kg of prednis(ol)one per day

Exclusion Criteria:

* Pregnant or lactating women
* A history of malignancy of any type, other than surgically excised non-melanoma skin cancers or in situ cervical cancer within 5 years before the day of dosing
* Use of immunologic response modifiers with the following periods prior to Day 1: 1 week: cyclophosphamide; 4 weeks: intravenous immunoglobulin, Kinaret (anakinra) and Enbrel (etanercept); 12 weeks: Remicade (infliximab), Humira (adalimumab), Simponi (golimumab), Orencia (abatacept), Actemra (tocilizumab), Cimzia (certolizumab), Cosentyx (secukinumab), plasmapheresis; 6 months: Rituxan/MabThera (rituximab), ofatumumab, any other anti-CD20 antibody, other long acting biologics
* More than 0.5 mg/kg of prednis(ol)one per day ("low dose corticosteroids") within the two weeks prior to Day 1
* Use of proton pump inhibitor drugs such as omeprazole and esomeprazole
* Has received any investigational drug (or is currently using an investigational device) within the 30 days before receiving the first dose of study medication, or at least 5 times the respective elimination half-life time (whichever is longer)
* History of drug abuse within the precious 12 months
* Alcoholism or excessive alcohol use, defined as regular consumption of more than approximately 3 standard drinks per day
* Refractory nausea and vomiting, malabsorption, external biliary shunt, significant bowel resection that would preclude adequate study drug absorption
* History of anorexia nervosa or periods of three months or more of low body weight in the past 5 years
* Donation of a unit or more of blood or blood products within 4 weeks prior to Day 1
* History of solid organ transplant
* History of epilepsy or other forms of seizures in the last 5 years
* Positive for screening for human immunodeficiency virus, hepatitis B (surface and core antibodies unrelated to vaccination), or hepatitis C (anti-HCV antibody confirmed with Hep C RNA)
* History of active or latent tuberculosis (TB) infection (must test negative using the QuantiFERON test to be eligible)
* History of serious infections requiring intravenous (by catheter that delivers antibiotics into your blood) treatment
* Live vaccine within 28 days prior to baseline or plan to receive one during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2020-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- Australia (3):
  - Premier Specialists, Kogarah, New South Wales
  - Sinclair Dermatology, East Melbourne, Victoria
  - Royal Melbourne, Dermatology Office, Melbourne, Victoria
- Croatia (2):
  - Clinical Hospital Osijek, Osijek
  - Klinichki Bolnicki Centar Zagreb, Zagreb
- France (2):
  - Hôpital Avicenne, Bobigny, Siene-Saint Denis
  - Rouen University Hospital, Rouen
- Greece (4):
  - University General Hospital of Ioannina, Ioannina, Ioannina
  - University Hospital of Larissa, Larissa, Thessaly
  - Hospital of Venereal and Skin Diseases A.Syggros, Athens
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Israel (2):
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 13 centers in 5 countries from 22 January 2016 to 10 January 2020.
Pre-assignment Details: A total of 69 patients were screened for the study (52 patients in Part A and 18* patients in Part B). Of these, 41 unique patients were enrolled in the study (27 patients in Part A and 15* patients in Part B). *One patient who completed Part A of the study and later relapsed was enrolled in Part B.
Groups:
- Part A: Open-label PRN1008, 12 weeks; 12 weeks follow-up
- Part B: Open-label PRN1008, 24 weeks; 4 weeks follow-up
Period: Part A: 24 Weeks
Arm/Group | Part A | Part B
Started | 27 | 0
Completed | 24 | 0
Not Completed | 3 | 0
Not completed — Adverse Event | 3 | 0
Period: Part B: 28 Weeks
Arm/Group | Part A | Part B
Started | 0 | 15 (One patient who completed Part A and later relapsed was enrolled in Part B.)
Completed | 0 | 14
Not Completed | 0 | 1
Not completed — Worsening of pemphigus | 0 | 1

BASELINE CHARACTERISTICS:
Population: One patient who completed Part A of the study and later relapsed was enrolled in Part B. Therefore baseline results of one patient are repeated in Part B and total patient number is 15.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 27 | 15 | 42
Age, Categorical [Count of Participants; unit: Participants] — Population: One patient who completed Part A of the study and later relapsed was enrolled in Part B.
  Participants
    Part A: number analyzed (Participants) | 27 | 0 | 27
    Part A: <=18 years | 0 | 0 | 0
    Part A: Between 18 and 65 years | 24 | 0 | 24
    Part A: >=65 years | 3 | 0 | 3
    Part B: number analyzed (Participants) | 0 | 15 | 15
    Part B: <=18 years | 0 | 0 | 0
    Part B: Between 18 and 65 years | 0 | 15 | 15
    Part B: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One patient who completed Part A of the study and later relapsed was enrolled in Part B.
  Participants
    Part A: number analyzed (Participants) | 27 | 0 | 27
    Part A: Female | 15 | 0 | 15
    Part A: Male | 12 | 0 | 12
    Part B: number analyzed (Participants) | 0 | 15 | 15
    Part B: Female | 0 | 7 | 7
    Part B: Male | 0 | 8 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One patient who completed Part A of the study and later relapsed was enrolled in Part B.
  Participants
    Part A: number analyzed (Participants) | 27 | 0 | 27
    Part A: American Indian or Alaska Native | 0 | 0 | 0
    Part A: Asian | 1 | 0 | 1
    Part A: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Part A: Black or African American | 0 | 0 | 0
    Part A: White | 22 | 0 | 22
    Part A: More than one race | 0 | 0 | 0
    Part A: Unknown or Not Reported | 4 | 0 | 4
    Part B: number analyzed (Participants) | 0 | 15 | 15
    Part B: American Indian or Alaska Native | 0 | 0 | 0
    Part B: Asian | 0 | 2 | 2
    Part B: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Part B: Black or African American | 0 | 0 | 0
    Part B: White | 0 | 8 | 8
    Part B: More than one race | 0 | 0 | 0
    Part B: Unknown or Not Reported | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) including clinically significant changes in physical examination, laboratory tests, and vital signs. An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. TEAEs were defined as AEs that developed or worsened or became serious during on-treatment phase that was defined as the time from the start of study drug up to study completion.
Time Frame: Part A: until 24 weeks and Part B: until 28 weeks
Population: Safety Analysis population: All patients who received at least 1 dose of rilzabrutinib; used for all safety analyses
Measure: Number; unit: percentage of participants
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
percentage of participants
  Any TEAE | 74.1 | 86.7
  Any serious TEAE | 11.1 | 0
  Any TEAE leading to treatment discontinuation | 11.1 | 0

2. Primary Outcome: Percentage of Participants Who Are Able to Achieve Control of Disease Activity (CDA) Within 4 Weeks of Starting PRN1008 Treatment Without the Need for Doses of Prednisone or Prednisolone >0.5 mg/kg
Description: CDA was defined as the time at which new lesions cease to form and established lesions begin to heal.
Time Frame: 4 weeks
Population: Intent-to-Treat (ITT) population: All patients who received at least 1 dose of rilzabrutinib
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part A: Open-label PRN1008, 12 weeks; 12 week follow-up
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
percentage of participants | 51.9 [31.9 to 71.3] | 60.0 [32.29 to 83.66]

3. Secondary Outcome: Percentage of Participants Able to Achieve Control of Disease Activity (CDA) Without Corticosteroids Within 4 Weeks
Description: CDA was defined as the time at which new lesions cease to form and established lesions begin to heal.
Time Frame: 4 weeks
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
percentage of participants | 11.1 [2.4 to 29.2] | 6.7 [0.17 to 31.95]

4. Secondary Outcome: Percentage of Participants Able to Achieve a Complete Response (CR) Without Corticosteroids
Description: CR was defined as complete healing of all lesions and the absence of new lesions.
Time Frame: Part A: 12 weeks treatment and Part B: 24 weeks treatment
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
percentage of participants | 0 | 0

5. Secondary Outcome: Percentage of Participants Able to Achieve Complete Remission (CR) Without the Need for Doses of Prednisone or Prednisolone of Greater Than 0.5mg/kg
Description: CR was defined as complete healing of all lesions and the absence of new lesions.
Time Frame: Part A: 12 weeks treatment and Part B: 24 weeks treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
percentage of participants | 14.8 [4.2 to 33.7] | 33.3 [11.82 to 61.62]

6. Secondary Outcome: Time to Control of Disease Activity (CDA)
Description: CDA was defined as the time at which new lesions cease to form and established lesions begin to heal. Kaplan-Meier estimate median time is reported.
Time Frame: Part A: until 24 weeks and Part B: until 28 weeks
Population: ITT
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
days | 33.0 [29.0 to 58.0] | 29.0 [15.0 to 34.0]

7. Secondary Outcome: Time to End of Consolidation Phase (ECP)
Description: ECP was defined as the time at which no new lesions have developed for minimum of 2 weeks, and approximately 80% of existing lesions have healed. The median time to ECP was based on Kaplan-Meier estimate which considered censoring at end of follow-up for patients who didn't have an event. A +/-3 days window for visits at Week 3 and 5, and +/-7 days window for visits at Week 9, 13, 17, 21, 25.
Time Frame: Part A: until 24 weeks and Part B: until 28 weeks
Population: ITT
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
days | 170.0 [95.0 to NA] — The upper CI was not estimable due to the insufficient number of patients with an ECP response. | 58.0 [48.0 to NA] — The upper CI was not estimable due to the insufficient number of patients with an ECP response.

8. Secondary Outcome: Time to Complete Remission (CR)
Description: CR was defined as complete healing of all lesions and the absence of new lesions.
Time Frame: Part A: until 24 weeks and Part B: until 28 weeks
Population: ITT
Measure: Median (80% Confidence Interval); unit: days
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
days | NA [NA to NA] — Less than 50% patients achieved CR. | NA [NA to NA] — Less than 50% patients achieved CR.

9. Secondary Outcome: Time to Relapse After PRN1008 Treatment Discontinuation
Description: Relapse was defined as appearance of ≥3 new lesions/month that do not heal spontaneously within 1 week, or by extension of established lesions, in a patient who has achieved disease control. The median time to relapse was based on Kaplan-Meier estimate which considered censoring at end of follow-up for patients who didn't have an event. A +/-3 days window for visits at Week 3 and 5, and +/-7 days window for visits at Week 9, 13, 17, 21, 25.
Time Frame: Part A: until 24 weeks and Part B: until 28 weeks
Population: ITT
Measure: Median (Full Range); unit: days
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
days | 96.0 [27.0 to 99.0] | 198.0 [41.0 to 209.0]

10. Secondary Outcome: Cumulative Corticosteroid Usage
Description: Cumulative corticosteroid usage
Time Frame: Part A: until 24 weeks and Part B: until 28 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
mg | 983.43 (827.676) | 2089.600 (1274.011)

11. Secondary Outcome: Percentage Change From Baseline in Pemphigus Disease Area Index (PDAI) Total Activity Scores
Description: The PDAI questionnaire has 2 components including activity and damage. The activity component consists of skin, scalp and mucosa parts, and the damage component consists of skin and scalp parts. The total activity score was used for the summary of PDAI scores. PDAI total activity score = Total skin activity + Total scalp activity + Total mucosa activity. PDAI Total Activity Score ranged from 0 to 250 points representing disease activity (higher scores mean a worse outcome). Negative change in total activity score from baseline indicates improvement in pemphigus activity.
Time Frame: Part A: until 24 weeks and Part B: until 28 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
score on a scale
  end of treatment: number analyzed (Participants) | 24 | 14
  end of treatment | -55.7 (40.91) | -78.60 (35.839)
  end of follow-up: number analyzed (Participants) | 24 | 14
  end of follow-up | -57.7 (38.45) | -59.68 (48.403)

12. Secondary Outcome: Change From Baseline in Autoimmune Bullous Skin Disorder Intensity Score (ABSIS) Total Activity Score
Description: ABSIS Total Activity Score ranged from 0 to 206 points representing disease activity (higher scores mean a worse outcome). Negative change in total activity score from baseline indicates improvement in pemphigus activity.
Time Frame: Part A: until 24 weeks and Part B: until 28 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
score on a scale
  end of treatment: number analyzed (Participants) | 24 | 14
  end of treatment | -8.18 (14.475) | -6.591 (4.7664)
  end of follow-up: number analyzed (Participants) | 24 | 14
  end of follow-up | -9.98 (18.369) | -5.705 (4.6248)

13. Secondary Outcome: Change From Baseline in Autoimmune Bullous Diseases Quality of Life (ABQOL)
Description: ABQOL score ranged from 0 to 68 points representing disease activity (higher scores mean a worse outcome).
Time Frame: Part A: until 24 weeks and Part B: until 28 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
score on a scale
  end of treatment: number analyzed (Participants) | 24 | 14
  end of treatment | -3.7 (6.96) | -6.36 (9.394)
  end of follow-up: number analyzed (Participants) | 24 | 14
  end of follow-up | -2.9 (6.71) | -3.79 (9.569)

14. Secondary Outcome: Change From Baseline in Treatment of Autoimmune Bullous Diseases Quality of Life (TABQOL) Scores
Description: TABQOL score ranged from 0 to 68 points representing disease activity (higher scores mean a worse outcome).
Time Frame: Part A: until 24 weeks and Part B: until 28 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
score on a scale
  end of treatment: number analyzed (Participants) | 24 | 14
  end of treatment | -0.0 (6.73) | -2.00 (6.051)
  end of follow-up: number analyzed (Participants) | 24 | 14
  end of follow-up | -0.1 (5.92) | -2.14 (5.655)

15. Secondary Outcome: Change From Baseline in Appetite (SNAQ Score)
Description: Simplified Nutritional Appetite Questionnaire (SNAQ) score ranged from 0 to 20 points representing disease activity (higher scores mean a better outcome).
Time Frame: Part A: until 24 weeks and Part B: until 28 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part A | Part B
Number analyzed (Participants) | 27 | 15
units on a scale
  end of treatment: number analyzed (Participants) | 24 | 14
  end of treatment | 1.1 (2.45) | 0.21 (2.082)
  end of follow-up: number analyzed (Participants) | 24 | 14
  end of follow-up | 1.0 (2.84) | 0.50 (2.103)

ADVERSE EVENTS:
Time Frame: Part A: until 24 weeks and Part B: until 28 weeks
Description: Reported AEs and deaths are TEAEs that developed, worsened, or became serious during the treatment period. Analysis was performed on safety population.
Arm/Group | Part A | Part B
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/15
Serious Adverse Events (participants affected / at risk) | 3/27 | 0/15
Other Adverse Events (participants affected / at risk) | 20/27 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (N=27) | Part B (N=15)
Pulmonary sequestration (Congenital, familial and genetic disorders) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (N=27) | Part B (N=15)
Nausea (Gastrointestinal disorders) | 6 | 4
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Staphylococcal skin infection (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Headache (Nervous system disorders) | 4 | 1
Dizziness (Nervous system disorders) | 2 | 2
Paraesthesia (Nervous system disorders) | 2 | 0
Fatigue (General disorders) | 2 | 1
Peripheral swelling (General disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Change of bowel habit (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Teeth brittle (Gastrointestinal disorders) | 0 | 1
Dermatophytosis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Androgenetic alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Asthenia (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Terminal insomnia (Psychiatric disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hot flush (Vascular disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT02704429/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT02704429/SAP_001.pdf